CLINICAL TRIAL: NCT01821404
Title: The Impact of Atorvastatin on Prostate Cancer - a Randomized, Pre-surgical Clinical Trial
Brief Title: Atorvastatin Before Prostatectomy and Prostate Cancer
Acronym: ESTO1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Fimlab laboratories (Unknown); University of Eastern Finland (Other); Finnish Cultural Foundation (Other)
Responsible Party: Principal Investigator, Teemu Murtola, Clinical teacher, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-005438-20
Record Dates: First submitted 2013-03-22; First posted 2013-04-01 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Prostatic Neoplasms
Keywords: Apoptosis; Atorvastatin; Inflammation; Pre-surgical trial; Proliferation; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Similar capsules as in the atorvastatin arm, but including no active ingredient. Used daily for 3-5 weeks before prostatectomy
  Interventions: Drug: Placebo
- Atorvastatin (Experimental): Atorvastatin capsules orally, 80 mg daily for 3-5 weeks before prostatectomy
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Capsules including 80 mg of atorvastatin
  Arms: Atorvastatin
Drug: Placebo — Similar capsules as in the atorvastatin arm, but without the active ingredient
  Arms: Placebo

SUMMARY:
This single-center, randomized, double-blind trial assesses the impact of short-term atorvastatin administration on proliferation activity, apoptotic rate and histological inflammation in prostate tissue.

DETAILED DESCRIPTION:
In this trial 160 men who have been diagnosed with prostate cancer, and whose first-line treatment will be radical prostatectomy (surgical removal of the prostate), are randomized to receive either 80 mg atorvastatin or placebo daily for 2-5 weeks until the operation. Blood cholesterol and serum PSA are measured before starting the study drug use and before the operation.

After the operation change in PSA and histological inflammation, apoptotic rate and Ki-67 staining intensity are compared between atorvastatin-treated and placebo-treated men. The correlation between changes in serum cholesterol or prostate specific antigen (PSA) and the tissue characteristics is evaluated.

After recruiting 60 men we will perform an interim analysis on primary end-points without breaking the blinding to treatment allocation. If we observe a statistically significant difference in all primary end-points, the trial will be stopped early and the results published.

Additionally, atorvastatin concentration in the blood and the prostate tissue is measured with mass spectrometry to determine penetrance of atorvastatin into the prostate. DNA- and RNA-samples are obtained from the prostate tissue and the blood. These will be used to study how gene expression of statin- and cholesterol-modifying enzymes affects the responses observed in prostate tissue.

As a secondary end-point we will measure recovery of erectile function after the operation and compare between the two study arms. Erectile function is measured using IIEF-5 questionnaire once before the operation and again 3, 6, 9 and 12 months from the prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer proven histologically in prostate biopsy
* Radical prostatectomy selected as the first-line treatment
* Willingness to participate and sign informed consent

Exclusion Criteria:

* Previous oncological treatments for any malignancy
* Previous usage of statins, finasteride or dutasteride within a year prior to prostate cancer diagnosis
* Clinically significant liver- or kidney insufficiency (plasma alanine aminotransferase level is twice over the recommended upper limit or serum creatinine level is over 170 µmol/l)
* Previous adverse effects from cholesterol-lowering treatment
* Ongoing use of drugs having interactions with statins (St John's Wort, HIV protease inhibitors, ciclosporin, macrolide antibiotics, fusidic acid, phenytoin, carbamazepine, dronedarone or oral antifungal medication)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Apoptosis | Four weeks after recruitment
  Number of apoptotic cells in prostate tissue. Measured after radical prostatectomy, on average after 4 weeks of recruitment
Ki-67 expression | Four weeks after recruitment
  Cellular proliferation activity in prostate tissue as measured by Ki-67 expression. Measured after radical prostatectomy, on average after 4 weeks of recruitment
Histological inflammation | After prostatectomy
  Extent of histological inflammation in the prostate tissue as evaluated by study pathologist
serum PSA | At recruitment and before prostatectomy
  Change in serum PSA level as measured before starting the study drug and again just before prostatectomy

SECONDARY OUTCOMES:
serum cholesterol | At recruitment and again four weeks after
  Changes in measured fasting serum cholesterol parameters: total cholesterol, HDL and LDL. First measure is done at recruitment, another right before radical prostatectomy.
Atorvastatin level in prostate tissue | Four weeks after recruitment
  Measurement of atorvastatin level in prostate tissue with mass spectrometry. Measured after radical prostatectomy, on average four weeks after recruitment

OTHER OUTCOMES:
Genotype of cholesterol-metabolizing enzymes | Post-hoc analysis, one year after recruitment completes
  Genotyping of cholesterol-metabolizing enzymes from blood and tissue samples
Genotype of statin-metabolizing enzymes | Post hoc analysis, one year after recruitment completes
  Genotyping statin-metabolizing enzymes from blood and tissue samples
Erection function | One year after prostatectomy
  Erectile function as measured with IIEF-5 questionnaire before prostatectomy and again at 3 month intervals during the first year after prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Teemu J Murtola, M.D., Ph.D., Principal Investigator — Tampere University; Teuvo LJ Tammela, M.D., Ph.D., Study Director — Tampere University
Locations (3):
- Finland (3):
  - Päijät-Häme Central Hospital, Lahti
  - Satakunta Central Hospital, Pori
  - Tampere University Hospital, Department of Urology, Tampere

REFERENCES:
- [Derived] Raittinen PVH, Syvala H, Tammela TLJ, Hakkinen MR, Ilmonen P, Auriola S, Murtola TJ. Atorvastatin induces adrenal androgen downshift in men with prostate cancer: A post Hoc analysis of a pilot adaptive Randomised clinical trial. EBioMedicine. 2021 Jun;68:103432. doi: 10.1016/j.ebiom.2021.103432. Epub 2021 Jun 16. PMID 34144486